CLINICAL TRIAL: NCT05507671
Title: The Role of the Bacillus Calmette-Guérin Vaccine (BCG) in the Clinical Evolution of COVID-19 and in the Efficacy of Anti-SARS-CoV-2 (Severe Acute Respiratory Syndrome Coronavirus 2) Vaccines
Brief Title: The Role of BCG Vaccine in the Clinical Evolution of COVID-19 and in the Efficacy of Anti-SARS-CoV-2 Vaccines
Acronym: SARS-CoV-2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Oswaldo Cruz Foundation (Other)
Collaborators: University of Sao Paulo (Other); Federal University of Juiz de Fora (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BCG-COVID/484016302711489/2020
Record Dates: First submitted 2021-05-27; First posted 2022-08-19 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-03

CONDITIONS: COVID-19
Keywords: COVID-19; SARS-CoV-2; BCG vaccine; Bacillus Calmette-Guérin; clinical trials; trained immunity
MeSH Terms: conditions — COVID-19 | interventions — Vaccines

STUDY DESIGN:
Intervention Model Description: Two-arm study, BCG vaccine versus placebo, to assess the effect of BCG in preventing severe form of covid19 and improving the efficacy of anti-SARS-CoV-2 vaccines
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not be informed if they received BCG or placebo. They will be informed that the injection may or may not give a local reaction regardless of what they receive.
  Blood samples for serological and cytokine studies will be coded and the laboratory technician will not know which samples are from participants who received BCG or placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BCG vaccine (Active Comparator): BCG (Bacillus Calmette-Guérin) vaccine - 0,1ml intradermal
  Interventions: Biological: BCG (Bacillus Calmette-Guérin) vaccine
- Placebo (Placebo Comparator): Solvent of BCG vaccine - 0,1ml intradermal
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: BCG (Bacillus Calmette-Guérin) vaccine — Application of BCG vaccine (0.1 ml intradermal) in the right arm deltoid insertion
  Arms: BCG vaccine
Other: Placebo — Application of BCG solvent (0.1 ml intradermal) in the right arm deltoid insertion
  Arms: Placebo

SUMMARY:
Clinical trial with randomized allocation in two arms (BCG vaccine versus placebo) of volunteers at risk but not yet infected nor vaccinated against SARS-CoV-2. Initially will be evaluated whether BCG has a protective role against severe form of the disease. After participants are vaccinated against COVID-19, it will be evaluated whether BCG favors the vaccine's efficacy. Volunteers will be recruited in three Brazilian states, with at least 250 seronegative in each group. The BCG-trained immunity stimulus will be investigated by assessing cytokines at D0 and D60 in a subsample of 50 participants per group. Until being vaccinated against COVID-19, the participants will be followed for up to 6 months, with visits scheduled every 2 months for interviews and immunoglobulin G (IgG) anti-SARS-CoV-2 antibodies. Those who become symptomatic at any time during the follow-up will be guided and monitored remotely daily until the end of their clinical evolution. After being vaccinated against COVID-19, visits to participants will be adjusted for the time of vaccination (VD), 20 days after the 1st dose (P1) and at least 30 days (P2) after the 2nd dose, with the aim of comparing the efficacy of the anti-SARS-CoV-2 vaccine in the two groups in the short and medium term.

The study's conclusions on the efficacy of BCG in preventing severe COVID-19 will be based on: incidence of SARS-Cov-2 infection (defined as the emergence of IgG over the follow-up period); incidence of illness by COVID-19 (defined as the presence of symptoms among infected participants); intensity and duration of symptoms between cases of COVID-19 and frequency and duration of hospitalizations for COVID-19 in each group. The occurrence, type, frequency and intensity of adverse effects associated with vaccination of adults with BCG will be reported.

The study's conclusions regarding the effect of BCG on efficacy of vaccines against COVID-19 will be based on: frequency of anti-SARS-CoV-2 neutralizing antibodies after the vaccine' 1st and 2nd doses in both groups.

DETAILED DESCRIPTION:
1. OBJECTIVE- To evaluate the role of the BCG vaccine against the severe form of COVID-19 and in improving the efficacy of anti-SARS-CoV-2 vaccines through a two-arm clinical trial comparing BCG versus placebo. Specifically:

   1. Assess whether BCG vaccine is able to stimulate the nonspecific immune response (trained immunity)
   2. Verify whether BCG is able to protect against SARS-CoV-2 infection
   3. Assess whether BCG is able to protect infected with SARS-CoV-2 against illness
   4. Assess whether BCG is able to protect subjects with COVID-19 against its severe form
   5. Evaluate whether BCG can favor the effectiveness of doses of anti-SARS-CoV-2 vaccines
   6. Knowing whether revaccination of adults with BCG causes unexpected adverse reactions
2. METHODOLOGY:

   2.1 STUDY MODEL: Two-arm Clinical Trial - intervention (BCG) versus placebo

   2.2 STUDY POPULATION: Volunteers not yet infected with SARS-CoV-2 or vaccinated against COVID-19, who can be essential service workers with frequent contact with the population: workers in health posts, users of the public health network due to others non-serious illnesses, police officers, employees of pharmacies, supermarkets, stores and others

   Sampling: As the real prevalence of SARS-CoV-2 infection in the eligible population of the different recruitment sites is unknown, a prevalence of 50% was considered (it provides the largest sample size) and estimated that the post-BCG prevalence would decrease at least 10% if its effectiveness to be demonstrated. Thus, it was found a sample of 385 subjects. Considering losses, a minimum of 400 participants will be recruited, with at least 200 in each group.

   2.3. INCLUSION CRITERIA:
   * Never been infected by SARS-Cov-2 - clinical history and absence of anti-SARS-CoV-2 immunoglobulins IgM/IgG antibodies by rapid test (immediate) and serology test (later confirmation)
   * Not having been vaccinated against COVID-19
   * Be at least 18 years old

   2.4. EXCLUSION CRITERIA: • Have been vaccinated with BCG less than 6 months ago

   • Have been vaccinated with BCG more than once in the past
   * Present any classic contraindications for BCG - pregnancy, breastfeeding, acute febrile illness, severe allergy to one of the components, vaccination with other live vaccines in the last month (measles, yellow fever, herpes zoster), immunosuppression for any cause (congenital, illness, use of corticosteroids or immunosuppressants)
   * Have had tuberculosis or contacted someone with tuberculosis
   * Present signs of any current acute illness or have had a severe illness less than 15 days
   * Present a skin lesion at the vaccine application site (right deltoid muscle)
   * History of severe allergic reactions to any product: urticaria, glottis edema, angioedema, respiratory failure, bronchospasm
   * History of serious autoimmune diseases: systemic lupus erythematosus, Crohn's disease, ulcerative colitis, multiple sclerosis, hemolytic anemia, ankylosing spondylitis, pemphigus and others
   * Immunocompromise for any reason: congenital, illness, use of corticosteroids or immunosuppressants
   * Presenting a risk comorbidity for severe COVID-19: poorly controlled hypertension, decompensated heart disease (chronic, congenital or ischemic), pulmonary disease (chronic pneumopathy, poorly controlled asthma, chronic interstitial pneumopathy, others ...), disease advanced chronic kidney disease (use of dialysis), transplantation (of solid organs or bone marrow), uncontrolled diabetes

   2.5. RECRUITMENT OF PARTICIPANTS The volunteers will be recruited in three different Brazilian states - Minas Gerais state (Juiz de Fora city), Amazonas state (Manaus city) and Pará state (Belém city). Their approach will be based on the viability and logistics of each recruitment site, considering the local dynamics of anti-COVID-19 vaccination by age. Those who meet the inclusion criteria and accept to participate in the study, must sign the Informed Consent Form (ICF). By lot, the participant will be allocated to Group 1 or 2, to receive placebo (BCG solvent) or BCG vaccine.

   2.6. INCLUSION AND FOLLOW-UP OF PARTICIPANTS 2.6.a -- Evaluation of BCG against the severe form of COVID-19:

   The subjects will be contacted at D0 (day of inclusion and intervention), D60, D120 and D180, as well as on any day of symptom onset in order to assess the presence and evolution of a SARS-CoV-2 infection. A standardized questionnaire will be developed and tablets will be programmed with the REDCap software to conduct interviews at each visit to investigate demographic data, past and current illnesses, vaccination history, risk activities and symptoms suggestive of COVID-19. Participants will be instructed to inform the team as soon as present any suspicious symptoms. In each scheduled visit, the participants will also undergo a venous blood collection to:

   - On D0 - Search of IgM/IgG antibodies by rapid test and IgG by serology (enzyme immunoassay-ELISA) in all subjects and search of pro-inflammatory cytokines Tumor Necrosis Factor α (TNF-α), interferon γ (IFN-γ), interleukin (IL)1β, IL-4, IL-6 and IL-10 in 50 participants from each group.

   - On D60 - Search of anti-SARS-CoV-2 IgG by ELISA in all participants and paired cytokine search (participants who did it on D0).
   * On D120 and D180 - Search of anti-SARS-CoV-2 IgG by ELISA.
   * If Symptom - Daily follow-up to guide diagnostic confirmation of SARS-CoV-2 infection in the local health network and to monitor clinical evolution. Furthermore, the patient will fill a table of daily symptoms, which will be collected at the next scheduled visit. In case of hospitalization, data of clinical evolution will be obtained from medical records.

   2.6.b -- Evaluation of BCG´s capacity to improve the vaccine anti-SARS-CoV-2 efficacy:

   From the moment the participants are vaccinated against covid-19, the visits will be adjusted to the vaccination schedule, as follows:

   - VD - at the time of 1st dose of the vaccine

   - P1 - 20 days after the 1st dose

   - P2 - at least 30 days after the 2nd dose On all these occasions, neutralizing anti-SARS-CoV-2 antibodies will be tested in all participants.

   2.7. INTERVENTION The inclusion in the BCG or Placebo Group will be done by lot, whose knowledge will be restricted to the main researcher and the professional who will perform the intervention. The participants and the technician who will carry out the laboratory tests will not know it.

   - BCG Group - BCG vaccine (live attenuated Mycobacterium bovis (Bacillus Calmette-Guérin) from the Serum Institute of India Ltd. Intradermal dose of 0.1 ml applied at the distal insertion of the right deltoid.

   Expected adverse effects of BCG can be tenderness, swelling and a reddened papule at the site which will become a 1 cm-diameter liquid ulcer that will close in 2 or 3 months, almost always leaving a scar of the same size. Other possible side effects are: headache, malaise, fever, ulcer greater than 1 cm, delayed healing (up to 6 months), enlarged lymph nodes. A rare serious complication is local or axillary node abscess due to error in administration with subcutaneous deposit of the vaccine. Thus, BCG will be managed by a rigorously trained professional. There is also reference to the spread of the vaccine bacillus causing organ damage in immunocompromised individuals (an exclusion criterion). Subjects with a severe reaction will receive adequate follow-up and treatment.

   -Placebo Group - Application of 0.1 ml intradermal of BCG vaccine solvent.

   2.8. INFECTION DETECTION Current SARS-Cov-2 infection will be identified by rapid test to detect IgM/IgG antibodies (only on D0 as an exclusion criterion) and by serology to detect IgG antibodies on every visit. Through positivity for IgG throughout the follow-up, the investigators will identify the participants who became infected between visits throughout the follow-up.

   2.9. CLINICAL EVOLUTION - The clinical status of symptomatic infected people will be defined as:
   * MILD STATUS (Influenza Syndrome-SG) - Fever accompanied by cough or sore throat or loss of smell/taste and at least one of the following symptoms: headache, myalgia or arthralgia. Less common symptoms may be: body pain, nasal congestion, diarrhea, abdominal pain, rash, discolored fingers and toes, conjunctivitis.
   * MODERATE STATUS - Tiredness or slight difficulty in breathing on small efforts and/or increase in the intensity of the underlying symptoms after 4 days of illness and/or increase in the number of underlying symptoms after 4 days of illness and/or persistence of symptoms for more than one week.
   * SERIOUS STATUS (Severe Acute Respiratory Syndrome) - SG associated with deficit in the respiratory system (difficulty breathing, cyanosis, oxygen saturation <95%, tachypnea, partial pressures of oxygen in alveolar gas/fraction of inspired oxygen (PaO2/FiO2) <300 and/or pulmonary infiltration >50% in 24- 48h), deficit in the cardiovascular system (hypotension, weak pulse) or change in mental status.
   * CRITICAL STATUS - Respiratory failure, septic shock and / or multiple organ dysfunction, loss of speech or movement.

   2.10. EVALUATION OF THE HUMORAL RESPONSE PROFILE At D0, as an inclusion criterion, the rapid test for detection of anti-SARS-CoV-2 IgG/IgM antibodies (TR COVID-19 IgM/IgG "BioManguinhos-Fiocruz") with 100% specificity for IgM and IgG and sensitivity of 85.7% (4-7 days) and 90% (> 8 days) for IgM and 92.8% (4-7 days) and 90% (>8 days) for IgG. Also on D0 and on all visiting days and in case of symptoms, IgG will be detected by a commercial enzyme immunoassay (recombinant ELISA - "Euroimmun Brasil Medicina Diagnóstica") with the S1 subdomain of the Spike protein as the capture antigen, in order to detect infections occurred between visits (seroconversion).

   To assess the efficacy of anti-SARS-CoV-2 vaccines, anti-SARS-CoV-2 neutralizing antibodies will be investigated using the SARS-CoV-2 Surrogate Virus Neutralization Test-sVNT ("Genscript") kit, which provides qualitative and semi-quatitative (titer in UI/ml) results. This investigation will be done 20 days after the 1st dose and at least 1 month after the 2nd dose of the vaccine.

   2.11. CYTOKINE ANALYSIS - It will be measure the proinflammatory cytokines IL-1β, IL-4, IL-6, IL-10, TNF-α (R&D Systems) and IFN-γ ("Sanquin") at D0 and D60 to assess the effectiveness of BCG in stimulating the non-specific immune response.

   2.12. ETHICAL ISSUES - The project was approved by the National Commission for Ethics in Research with Human Beings-CONEP. Volunteers who wished to participate signed the Informed Consent Form. An Independent Data and Safety Monitoring Committee (IDSMC) will monitor the study to ensure it is ethically non-violent and data credible, and may recommend modifications or suspension of the study if necessary. Through the Research Electronic Data Capture-REDCap software, a data manager will provide information about the study progress any time it be requested. The results of the exams will be provided to the participants. Intense reaction to BCG will receive due care from the research team and will be notified to CONEP and IDSMC within 24 hours. Participants will be encouraged to receive the COVID-19 vaccine when it becomes available to them.

   2.14. STATISTICAL ANALYSIS OF RESULTS - Through the Statistical Package for the Social Sciences (IBM SPSS v.22) and Stata (v.14.0) programs, the outcomes will be analyzed comparatively between the groups, being defined as failures. Analyzes will be performed for the intention-to-treat population (total recruits) and per protocol population (with full follow-up) using the Kaplan-Meier method. Proportions will be calculated with 95% confidence intervals and compared by Chi2 and Fisher's exact test. Survival curves will be compared by log rank test. Logistic regression will identify the set of independent variables that can explain the binary dependent variables, such as serological reactivity.

ELIGIBILITY:
INCLUSION CRITERIA:

* Never been infected by SARS-Cov-2 - clinical history and absence of anti-SARS-CoV-2 IgM/IgG antibodies by the rapid test (immediate) and by serology test (later confirmation)
* Not having been vaccinated against COVID-19
* Be at least 18 years old

EXCLUSION CRITERIA:

* Have been vaccinated with BCG less than 6 months ago
* Have been vaccinated with BCG more than once in the past
* Present any classic contraindications for BCG - pregnancy, breastfeeding, acute febrile illness, severe allergy to one of the components, vaccination with other live vaccines in the last month (measles, yellow fever, herpes zoster), immunosuppression for any cause (congenital, illness, use of corticosteroids or immunosuppressants)
* Have had tuberculosis or contacted someone with tuberculosis
* Present signs of any current acute illness or have had a severe illness less than 15 days
* Present a skin lesion at the vaccine application site (right deltoid muscle)
* History of severe allergic reactions to any product: urticaria, glottis edema, angioedema, respiratory failure, bronchospasm
* History of serious autoimmune diseases: systemic lupus erythematosus, Crohn's disease, ulcerative colitis, multiple sclerosis, hemolytic anemia, ankylosing spondylitis, pemphigus and others
* Immunocompromise for any reason (congenital, illness, use of corticosteroids or immunosuppressants)
* Presenting a risk comorbidity for severe COVID-19, such as: poorly controlled hypertension, decompensated heart disease (chronic, congenital or ischemic), pulmonary disease (chronic pneumopathy, poorly controlled asthma, chronic interstitial pneumopathy, others ...), disease advanced chronic kidney disease (use of dialysis), transplantation (of solid organs or bone marrow), uncontrolled diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 556 (Estimated)
Dates: Start 2021-05-27 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of SARS-Cov-2 infection in both groups over the follow-up | Up to six months from recruitment day
  Appearance of IgG antibodies (seroconversion) in the participants not yet vaccinated against COVID-19
Incidence of illness by COVID-19 in both groups over the follow-up | Up to six months from recruitment day
  Presence of symptoms among subjects not vaccinated against COVID-19 diagnosed with infection after D0 or seroconverted
Intensity of the efficacy of the first dose of the vaccine against COVID-19 | Up to six months from recruitment day
  Comparison of groups regarding frequency and titer (UI/ml) of anti-SARS-CoV-2 neutralizing antibodies after first dose of the specific vaccine, through the qualitative and semi-quatitative "SARS-CoV-2 Surrogate Virus Neutralization Test (sVNT)" Genscript Kit
Duration of the efficacy of the second dose of the vaccine against COVID-19 | One year from recruitment day
  Comparison of groups regarding frequency and titer (UI/ml) of anti-SARS-CoV-2 neutralizing antibodies after second dose of the specific vaccine, through the qualitative and semi-quatitative "SARS-CoV-2 Surrogate Virus Neutralization Test (sVNT)" Genscript Kit

SECONDARY OUTCOMES:
Intensity of clinical presentation of SARS-CoV-2 infection in both groups over the follow-up | One year from recruitment day
  Comparison of groups regarding the frequency of infected with mild, moderate, serious or critical symptoms (according to detailed description in item 2.9-Clinical Evolution) and deaths by COVID-19 during the follow-up. The information will be obtained through daily telephone interview, self-completion of a questionnaire and hospitalization data.
Duration of symptoms among participants with COVID-19 | Six months from recruitment day
  Comparison of groups regarding the duration (number of days) of symptoms among participants who acquire COVID-19. The information will be obtained through daily telephone interview, self-completion of a questionnaire and hospitalization data
Serum levels of cytokines after BCG vaccine stimulus (Trained Immunity effect) | Two months from recruitment day
  Comparison of serum concentrations (pg/mL) of cytokines TNF-α, IFN-γ, IL-1β, IL-4, IL-6 and IL-10 at D0 versus D60 of 50 participants of BCG group compared to 50 participants of placebo group

OTHER OUTCOMES:
Adverse effects correlated with BCG vaccine in adults | Six months from recruitment day
  Occurrence, type, frequency and intensity of adverse effects correlated with BCG revaccination obtained from obtained by interviewing those vaccinated with BCG (descriptive data)

CONTACTS AND LOCATIONS:
Overall Officials: Simone Ladeia-Andrade, MD PhD, Principal Investigator — Oswaldo Cruz Institute, Oswaldo Cruz Foundation; Igor C Johansen, PhD, Study Chair — University of Campinas, Brazil; Marcelo U Ferreira, MD PhD, Study Chair — University of Sao Paulo; Kezia KG Scopel, PhD, Study Chair — Universidade Federal de Juiz de Fora; Helena LC Santos, PhD, Study Chair — Oswaldo Cruz Institute, Oswaldo Cruz Foundation; Haroldo J Matos, MD PhD, Study Chair — Centro Universitário do Pará; Irineide A Antunes, MD, Study Chair — Policlínica Cardoso Fontes de Manaus; Lucilaide O Santos, MD, Study Chair — Fundação de Medicina Tropical Doutor Heitor Vieira Dourado; Sandra HC Tibiriça, MD PhD, Study Chair — Universidade Federal de Juiz de Fora
Locations (4):
- Brazil (4):
  - Policlínica Cardoso Fontes, Manaus, Amazonas
  - Universidade Federal de Juiz de Fora, Juiz de Fora, Minas Gerais
  - Centro Universitário do Pará, Belém, Pará
  - Oswaldo Cruz Foundation, Rio de Janeiro, Rio de Janeiro

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu F, Zhao S, Yu B, Chen YM, Wang W, Song ZG, Hu Y, Tao ZW, Tian JH, Pei YY, Yuan ML, Zhang YL, Dai FH, Liu Y, Wang QM, Zheng JJ, Xu L, Holmes EC, Zhang YZ. A new coronavirus associated with human respiratory disease in China. Nature. 2020 Mar;579(7798):265-269. doi: 10.1038/s41586-020-2008-3. Epub 2020 Feb 3. PMID 32015508
- [Background] Pan Y, Zhang D, Yang P, Poon LLM, Wang Q. Viral load of SARS-CoV-2 in clinical samples. Lancet Infect Dis. 2020 Apr;20(4):411-412. doi: 10.1016/S1473-3099(20)30113-4. Epub 2020 Feb 24. No abstract available. PMID 32105638
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Zhao J, Yuan Q, Wang H, Liu W, Liao X, Su Y, Wang X, Yuan J, Li T, Li J, Qian S, Hong C, Wang F, Liu Y, Wang Z, He Q, Li Z, He B, Zhang T, Fu Y, Ge S, Liu L, Zhang J, Xia N, Zhang Z. Antibody Responses to SARS-CoV-2 in Patients With Novel Coronavirus Disease 2019. Clin Infect Dis. 2020 Nov 19;71(16):2027-2034. doi: 10.1093/cid/ciaa344. PMID 32221519
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Corman VM, Landt O, Kaiser M, Molenkamp R, Meijer A, Chu DK, Bleicker T, Brunink S, Schneider J, Schmidt ML, Mulders DG, Haagmans BL, van der Veer B, van den Brink S, Wijsman L, Goderski G, Romette JL, Ellis J, Zambon M, Peiris M, Goossens H, Reusken C, Koopmans MP, Drosten C. Detection of 2019 novel coronavirus (2019-nCoV) by real-time RT-PCR. Euro Surveill. 2020 Jan;25(3):2000045. doi: 10.2807/1560-7917.ES.2020.25.3.2000045. PMID 31992387
- [Background] Gates B. Responding to Covid-19 - A Once-in-a-Century Pandemic? N Engl J Med. 2020 Apr 30;382(18):1677-1679. doi: 10.1056/NEJMp2003762. Epub 2020 Feb 28. No abstract available. PMID 32109012
- [Background] Hopman J, Allegranzi B, Mehtar S. Managing COVID-19 in Low- and Middle-Income Countries. JAMA. 2020 Apr 28;323(16):1549-1550. doi: 10.1001/jama.2020.4169. No abstract available. PMID 32176764
- [Background] Wang M, Cao R, Zhang L, Yang X, Liu J, Xu M, Shi Z, Hu Z, Zhong W, Xiao G. Remdesivir and chloroquine effectively inhibit the recently emerged novel coronavirus (2019-nCoV) in vitro. Cell Res. 2020 Mar;30(3):269-271. doi: 10.1038/s41422-020-0282-0. Epub 2020 Feb 4. No abstract available. PMID 32020029
- [Background] Gautret P, Lagier JC, Parola P, Hoang VT, Meddeb L, Mailhe M, Doudier B, Courjon J, Giordanengo V, Vieira VE, Tissot Dupont H, Honore S, Colson P, Chabriere E, La Scola B, Rolain JM, Brouqui P, Raoult D. RETRACTED: Hydroxychloroquine and azithromycin as a treatment of COVID-19: results of an open-label non-randomized clinical trial. Int J Antimicrob Agents. 2020 Jul;56(1):105949. doi: 10.1016/j.ijantimicag.2020.105949. Epub 2020 Mar 20. PMID 32205204
- [Background] Mahase E. Covid-19: what treatments are being investigated? BMJ. 2020 Mar 26;368:m1252. doi: 10.1136/bmj.m1252. No abstract available. PMID 32217607
- [Background] Colditz GA, Berkey CS, Mosteller F, Brewer TF, Wilson ME, Burdick E, Fineberg HV. The efficacy of bacillus Calmette-Guerin vaccination of newborns and infants in the prevention of tuberculosis: meta-analyses of the published literature. Pediatrics. 1995 Jul;96(1 Pt 1):29-35. PMID 7596718
- [Background] Mangtani P, Abubakar I, Ariti C, Beynon R, Pimpin L, Fine PE, Rodrigues LC, Smith PG, Lipman M, Whiting PF, Sterne JA. Protection by BCG vaccine against tuberculosis: a systematic review of randomized controlled trials. Clin Infect Dis. 2014 Feb;58(4):470-80. doi: 10.1093/cid/cit790. Epub 2013 Dec 13. PMID 24336911
- [Background] Dye C. Making wider use of the world's most widely used vaccine: Bacille Calmette-Guerin revaccination reconsidered. J R Soc Interface. 2013 Jul 31;10(87):20130365. doi: 10.1098/rsif.2013.0365. Print 2013 Oct 6. PMID 23904584
- [Background] Arts RJW, Moorlag SJCFM, Novakovic B, Li Y, Wang SY, Oosting M, Kumar V, Xavier RJ, Wijmenga C, Joosten LAB, Reusken CBEM, Benn CS, Aaby P, Koopmans MP, Stunnenberg HG, van Crevel R, Netea MG. BCG Vaccination Protects against Experimental Viral Infection in Humans through the Induction of Cytokines Associated with Trained Immunity. Cell Host Microbe. 2018 Jan 10;23(1):89-100.e5. doi: 10.1016/j.chom.2017.12.010. PMID 29324233
- [Background] Covian C, Fernandez-Fierro A, Retamal-Diaz A, Diaz FE, Vasquez AE, Lay MK, Riedel CA, Gonzalez PA, Bueno SM, Kalergis AM. BCG-Induced Cross-Protection and Development of Trained Immunity: Implication for Vaccine Design. Front Immunol. 2019 Nov 29;10:2806. doi: 10.3389/fimmu.2019.02806. eCollection 2019. PMID 31849980
- [Background] Higgins JP, Soares-Weiser K, Lopez-Lopez JA, Kakourou A, Chaplin K, Christensen H, Martin NK, Sterne JA, Reingold AL. Association of BCG, DTP, and measles containing vaccines with childhood mortality: systematic review. BMJ. 2016 Oct 13;355:i5170. doi: 10.1136/bmj.i5170. PMID 27737834
- [Background] Biering-Sorensen S, Aaby P, Lund N, Monteiro I, Jensen KJ, Eriksen HB, Schaltz-Buchholzer F, Jorgensen ASP, Rodrigues A, Fisker AB, Benn CS. Early BCG-Denmark and Neonatal Mortality Among Infants Weighing <2500 g: A Randomized Controlled Trial. Clin Infect Dis. 2017 Oct 1;65(7):1183-1190. doi: 10.1093/cid/cix525. PMID 29579158
- [Background] Schaltz-Buchholzer F, Biering-Sorensen S, Lund N, Monteiro I, Umbasse P, Fisker AB, Andersen A, Rodrigues A, Aaby P, Benn CS. Early BCG Vaccination, Hospitalizations, and Hospital Deaths: Analysis of a Secondary Outcome in 3 Randomized Trials from Guinea-Bissau. J Infect Dis. 2019 Jan 29;219(4):624-632. doi: 10.1093/infdis/jiy544. PMID 30239767
- [Background] Hollm-Delgado MG, Stuart EA, Black RE. Acute lower respiratory infection among Bacille Calmette-Guerin (BCG)-vaccinated children. Pediatrics. 2014 Jan;133(1):e73-81. doi: 10.1542/peds.2013-2218. Epub 2013 Dec 30. PMID 24379224
- [Background] Nemes E, Geldenhuys H, Rozot V, Rutkowski KT, Ratangee F, Bilek N, Mabwe S, Makhethe L, Erasmus M, Toefy A, Mulenga H, Hanekom WA, Self SG, Bekker LG, Ryall R, Gurunathan S, DiazGranados CA, Andersen P, Kromann I, Evans T, Ellis RD, Landry B, Hokey DA, Hopkins R, Ginsberg AM, Scriba TJ, Hatherill M; C-040-404 Study Team. Prevention of M. tuberculosis Infection with H4:IC31 Vaccine or BCG Revaccination. N Engl J Med. 2018 Jul 12;379(2):138-149. doi: 10.1056/NEJMoa1714021. PMID 29996082
- [Background] deKernion JB, Golub SH, Gupta RK, Silverstein M, Morton DL. Successful transurethral intralesional BCG therapy of a bladder melanoma. Cancer. 1975 Nov;36(5):1662-7. doi: 10.1002/1097-0142(197511)36:53.0.co;2-6. PMID 1192356
- [Background] Wardhana, Datau EA, Sultana A, Mandang VV, Jim E. The efficacy of Bacillus Calmette-Guerin vaccinations for the prevention of acute upper respiratory tract infection in the elderly. Acta Med Indones. 2011 Jul;43(3):185-90. PMID 21979284
- [Background] Aiello A, Farzaneh F, Candore G, Caruso C, Davinelli S, Gambino CM, Ligotti ME, Zareian N, Accardi G. Immunosenescence and Its Hallmarks: How to Oppose Aging Strategically? A Review of Potential Options for Therapeutic Intervention. Front Immunol. 2019 Sep 25;10:2247. doi: 10.3389/fimmu.2019.02247. eCollection 2019. PMID 31608061
- [Background] Benn CS, Fisker AB, Whittle HC, Aaby P. Revaccination with Live Attenuated Vaccines Confer Additional Beneficial Nonspecific Effects on Overall Survival: A Review. EBioMedicine. 2016 Aug;10:312-7. doi: 10.1016/j.ebiom.2016.07.016. Epub 2016 Jul 15. PMID 27498365
- [Background] Roth AE, Benn CS, Ravn H, Rodrigues A, Lisse IM, Yazdanbakhsh M, Whittle H, Aaby P. Effect of revaccination with BCG in early childhood on mortality: randomised trial in Guinea-Bissau. BMJ. 2010 Mar 15;340:c671. doi: 10.1136/bmj.c671. PMID 20231251
- [Background] SERGENT E, CATANEI A, DUCROS-ROUGEBIEF H. [Antituberculous premunition by BCG; campaign followed from 1935 on 21,244 vaccinated and 20,063 non-vaccinated newborn infants; preliminary note]. Arch Inst Pasteur Alger. 1954 Mar;32(1):1-8. No abstract available. Undetermined Language. PMID 13181526
- [Background] Bricks LF. [Percutaneous or intradermal BCG vaccine?]. J Pediatr (Rio J). 2004 Mar-Apr;80(2):93-8. Portuguese. PMID 15079177
- [Background] Hoft DF, Leonardi C, Milligan T, Nahass GT, Kemp B, Cook S, Tennant J, Carey M. Clinical reactogenicity of intradermal bacille Calmette-Guerin vaccination. Clin Infect Dis. 1999 Apr;28(4):785-90. doi: 10.1086/515201. PMID 10825039
- [Background] Hesseling AC, Marais BJ, Gie RP, Schaaf HS, Fine PE, Godfrey-Faussett P, Beyers N. The risk of disseminated Bacille Calmette-Guerin (BCG) disease in HIV-infected children. Vaccine. 2007 Jan 2;25(1):14-8. doi: 10.1016/j.vaccine.2006.07.020. Epub 2006 Aug 1. PMID 16959383
- [Background] Baily GV. Tuberculosis prevention Trial, Madras. Indian J Med Res. 1980 Jul;72 Suppl:1-74. No abstract available. PMID 7005086
- [Background] Hatherill M, Geldenhuys H, Pienaar B, Suliman S, Chheng P, Debanne SM, Hoft DF, Boom WH, Hanekom WA, Johnson JL. Safety and reactogenicity of BCG revaccination with isoniazid pretreatment in TST positive adults. Vaccine. 2014 Jun 30;32(31):3982-8. doi: 10.1016/j.vaccine.2014.04.084. Epub 2014 May 9. PMID 24814553
- [Background] Buffen K, Oosting M, Quintin J, Ng A, Kleinnijenhuis J, Kumar V, van de Vosse E, Wijmenga C, van Crevel R, Oosterwijk E, Grotenhuis AJ, Vermeulen SH, Kiemeney LA, van de Veerdonk FL, Chamilos G, Xavier RJ, van der Meer JW, Netea MG, Joosten LA. Autophagy controls BCG-induced trained immunity and the response to intravesical BCG therapy for bladder cancer. PLoS Pathog. 2014 Oct 30;10(10):e1004485. doi: 10.1371/journal.ppat.1004485. eCollection 2014 Oct. PMID 25356988
- [Background] Escobar LE, Molina-Cruz A, Barillas-Mury C. BCG vaccine protection from severe coronavirus disease 2019 (COVID-19). Proc Natl Acad Sci U S A. 2020 Jul 28;117(30):17720-17726. doi: 10.1073/pnas.2008410117. Epub 2020 Jul 9. PMID 32647056
- [Background] Hegarty PK, Sfakianos JP, Giannarini G, DiNardo AR, Kamat AM. COVID-19 and Bacillus Calmette-Guerin: What is the Link? Eur Urol Oncol. 2020 Jun;3(3):259-261. doi: 10.1016/j.euo.2020.04.001. Epub 2020 Apr 13. PMID 32327396
- [Background] de Freitas E Silva R, Pitzurra R. What are the factors influencing the COVID-19 outbreak in Latin America? Travel Med Infect Dis. 2020 May-Jun;35:101667. doi: 10.1016/j.tmaid.2020.101667. Epub 2020 Apr 11. No abstract available. PMID 32289549
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Bolke E, Matuschek C, Fischer JC. Loss of Anti-SARS-CoV-2 Antibodies in Mild Covid-19. N Engl J Med. 2020 Oct 22;383(17):1694-1695. doi: 10.1056/NEJMc2027051. Epub 2020 Sep 23. No abstract available. PMID 32966710
- [Background] Wajnberg A, Amanat F, Firpo A, Altman DR, Bailey MJ, Mansour M, McMahon M, Meade P, Mendu DR, Muellers K, Stadlbauer D, Stone K, Strohmeier S, Simon V, Aberg J, Reich DL, Krammer F, Cordon-Cardo C. Robust neutralizing antibodies to SARS-CoV-2 infection persist for months. Science. 2020 Dec 4;370(6521):1227-1230. doi: 10.1126/science.abd7728. Epub 2020 Oct 28. PMID 33115920
- See also: Coronavirus World Health Organization (WHO) data — https://www.who.int/emergencies/diseases/novel-coronavirus-2019
- See also: Coronavirus data — https://www.who.int/emergencies/diseases/novel-coronavirus-2019?gclid=Cj0KCQiA962BBhCzARIsAIpWEL2M_wNxmazwA5Y4Ns6G3NNzIq6UICfkofpZuqjFd2UJ0qWFgDxH_ZQaAjNUEALw_wcB
- See also: Cases of coronavirus in Brazil — https://covid.saude.gov.br/
- See also: Number of coronavirus cases in Brazil — https://www.em.com.br/app/noticia/nacional/2020/04/16/interna_nacional,1139250/numero-de-casos-de-coronavirus-no-brasil-e-15-vezes-maior.shtml
- See also: COVID in young people — https://brasil.elpais.com/sociedade/2020-04-16/jovens-internados-mostram-rejuvenescimento-da-covid-19-no-brasil.html
- See also: Respiratory syndrome — https://www.msdmanuals.com/pt/profissional/doen%C3%A7as-infecciosas/v%C3%ADrus-respirat%C3%B3rios/coronav%C3%ADrus-e-s%C3%ADndromes-respirat%C3%B3rias-agudas-covid-19,-mers-e-sars
- See also: Novel coronavirus in suspected human cases — https://www.who.int/publications/i/item/10665-331501
- See also: Novel Coronavirus (2019-nCoV) Reverse Transcription Polymerase Chain Reaction (RT-PCR) Diagnostic Panel — https://www.fda.gov/media/134922/download
- See also: COVID-19 epidemiological bulletin — https://static.poder360.com.br/2020/05/boletim-epidemiologico-covid19-8mai2020-1.pdf
- See also: COVID-19: protecting health-care workers — https://doi.org/10.1016/S0140-6736(20)30644-9
- See also: Repositioning Chloroquine as Ideal Antiviral Prophylactic against COVID-19 - Time is Now — https://doi.org/10.1016/j.drudis.2020.06.030
- See also: Bacillus Calmette-guérin Vaccination to Prevent Infections of the Elderly — https://clinicaltrials.gov/ct2/show/record/NCT03296423
- See also: Leprosy prevention and control measures — https://www.saude.gov.br/saude-de-a-z/hanseniase/medidas-de-prevencao-e-controle
- See also: Correlation between universal BCG vaccination policy and reduced morbidity and mortality for COVID-19: an epidemiological study — https://www.medrxiv.org/content/10.1101/2020.03.24.20042937v2
- See also: Bacille Calmette-Guérin (BCG) vaccination and COVID-19 — https://www.who.int/news-room/commentaries/detail/bacille-calmette-guérin-(bcg)-vaccination-and-covid-19
- See also: BCG is a Good Immunotherapeutic Agent for Viral and Autoimmune Diseases: Is it a new weapon against coronavirus (COVID-19)? — https://www.ejgm.co.uk/article/bcg-is-a-good-immunotherapeutic-agent-for-viral-and-autoimmune-diseases-is-it-a-new-weapon-against-7892
- See also: BCG Vaccination to Protect Healthcare Workers Against COVID-19 — https://clinicaltrials.gov/ct2/show/NCT04327206
- See also: Reducing Health Care Workers Absenteeism in COVID-19 Pandemic Through BCG Vaccine (BCG-CORONA) — https://clinicaltrials.gov/ct2/show/NCT04328441
- See also: Vaccines available — https://familia.sbim.org.br/vacinas/vacinas-disponiveis/vacina-bcg
- See also: Normative Instruction Vaccination Calendar — https://www.saude.gov.br/images/pdf/2019/marco/22/Instrucao-Normativa-Calendario-Vacinacao-Site.pdf
- See also: BCG vaccine — https://www.ssi.dk/vaccinationer/vaccineleksikon/b/bcgvaccine-aj-vaccines
- See also: Consolidated Headquarters of the Ministry of Health of Brazil — https://bvsms.saude.gov.br/bvs/saudelegis/gm/2017/MatrizesConsolidacao/comum/240309.html
- See also: Intradermal vaccination against tuberculosis — https://www.ssi.dk/vaccinationer/injektionsteknik/intradermal-injektion-mod-tuberkulose
- See also: Coronavirus Clinical Management Protocol (COVID-19) in Primary Health Care. Version 02, March 2020, Ministry of Health of Brazil — https://www.saude.gov.br/images/pdf/2020/marco/20/20200318-ProtocoloManejo-ver002.pdf
- See also: Coronavirus — https://www.who.int/publications/i/item/10665-331501
- See also: SARS-CoV-2 specific antibody responses in COVID-19 patients — https://www.medrxiv.org/content/10.1101/2020.03.18.20038059v1
- See also: coronavirus Brazilian boletim — http://www.gov.br/saude/pt-br/centrais-de-conteudo/publicacoes/boletins/boletins-epidemiologicos/covid-19